CLINICAL TRIAL: NCT01594944
Title: Fetal Orbital Measurements by 3D Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC110046CTIL
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Orbital Volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will measure fetal orbital transverse and anterior-posterior diameter by 2D ultrasound and orbital volume by 3D ultrasound in women visiting our unit for other examinations during pregnancy. The investigators will examine 5-10 women in each gestational age in order to create a normal values curve throughout pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* well dated singleton pregnancies

Exclusion Criteria:

* multiple pregnancy
* pregnancies with known malformations,
* chromosomal abnormalities or
* intrauterine infections

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women 13-37w
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-05